CLINICAL TRIAL: NCT00236431
Title: A Randomized Double-Blind Placebo-Controlled Trial to Evaluate the Efficacy and Safety of Galantamine in Patients With Mild Cognitive Impairment (MCI) Clinically at Risk for Development of Clinically Probable Alzheimer's Disease
Brief Title: A Study to Evaluate the Efficacy and Safety of Galantamine in Patients With Mild Cognitive Impairment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR002014
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2010-11

CONDITIONS: Dementia; Alzheimer Disease
Keywords: Mild cognitive impairment; Galantamine hydrobromide; Memory disorders
MeSH Terms: conditions — Dementia; Alzheimer Disease; Cognitive Dysfunction; Memory Disorders | interventions — Galantamine

INTERVENTIONS:
Drug: Galantamine hydrobromide

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of galantamine treatment in patients with mild cognitive impairment.

DETAILED DESCRIPTION:
This is an international, multicenter, double-blind, randomized, placebo-controlled trial. Patients with mild cognitive impairment (MCI) who are clinically at risk for development of Alzheimer's disease will be treated for 24 months with either placebo or galantamine hydrobromide. Memory and overall clinical improvement will be evaluated using the Alzheimer's Disease Assessment Scale with cognitive subscale adapted to MCI (ADAS-cog/MCI) and the Clinical Dementia Rating Sum of the Boxes (CDR-SB). Overall functional skills and the severity of dementia will be assessed with the Clinical Dementia Rating Sum of the Boxes (CDR-SB) and the overall Clinical Dementia Rating (CDR) score. Additional assessments include the Digit Symbol Substitution Test (DSST) to measure attention. Safety will be assessed using adverse event reports, vital signs, laboratory parameters, physical examination, and electrocardiogram. The study hypothesis is that treatment with galantamine will be well tolerated and, compared with placebo, will significantly improve the signs and symptoms associated with mild cognitive impairment in patients who are considered likely to develop Alzheimer's disease. Galantamine hydrobromide immediate-release tablets (4, 8, or 12 milligrams), taken by mouth 2 times daily: 8mg/day for 4 weeks, 16mg/day for 4 weeks, then increased to 24mg/day for the remainder of the 24-month trial. Doses may be reduced at investigator's discretion after 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Clinical decline of cognitive ability consistent with mild cognitive impairment
* Delayed recall score <= 10 on a New York University paragraph recall test
* Sufficient visual, hearing and communication capabilities and be willing to complete serial standard tests of cognitive function
* Have a consistent informant to accompany them on scheduled visits
* Be able to read, write and fully understand the language of the cognitive scales used in the study

Exclusion Criteria:

* Neurodegenerative disorders such as Parkinson's disease
* Cognitive impairment resulting from acute cerebral trauma, hypoxic cerebral damage, vitamin deficiency states, infections such as meningitis or AIDS, or primary or metastatic cerebral neoplasia
* Epilepsy
* Significant psychiatric disease
* Peptic ulcer disease
* Clinically significant heart, lung, liver or kidney diseases
* Pregnant or nursing women or those without adequate contraception

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1063 (Actual)
Dates: Start 2001-05; Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Memory and cognition (ADAS-COG/MCI and CDR-SB scores), global functional skills and overall severity of dementia (the CDR-SB and the overall Clinical Dementia Rating) measured at 12 and 24 months.

SECONDARY OUTCOMES:
Digit Symbol Coding and Alzheimer's Disease Cooperative Study-ADL scale (MCI version) at 12 and 24 months. Safety assessment (reports of adverse events, laboratory values, results of physical examinations, and electrocardiograms) throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Lim AWY, Schneider L, Loy C. Galantamine for dementia due to Alzheimer's disease and mild cognitive impairment. Cochrane Database Syst Rev. 2024 Nov 5;11(11):CD001747. doi: 10.1002/14651858.CD001747.pub4. PMID 39498781
- See also: A study to evaluate the efficacy and safety of galantamine in patients with mild cognitive impairment. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=448&filename=CR002014_CSR.pdf